CLINICAL TRIAL: NCT00797784
Title: A Phase 2 Open Label Study to Assess the Efficacy and Safety of Etanercept (Enbrel®)for the Treatment of Discoid Lupus Erythematosus
Brief Title: The Safety and Efficacy of Etanercept (Enbrel®) for the Treatment of Discoid Lupus Erythematosus
Acronym: DISCLUP2008
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Academic Dermatology Centers (Other)
Responsible Party: Francisco A Kerdel,M.D., Florida Academic Dermatology Centers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FADC
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2008-11

CONDITIONS: Discoid Lupus Erythematosus (DLE)
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: etanercept(Enbrel®) — etanercept(Enbrel®) 50mgs subcutaneous (SC) injections twice weekly for 20 weeks

SUMMARY:
A 20 week study to assess the safety and efficacy of etanercept(Enbrel®)for the treatment of Discoid Lupus Erythematosus

ELIGIBILITY:
Inclusion Criteria:

* Subjects with discoid lupus erythematosus .Subjects require to have confirmation of diagnosis by a skin biopsy .This can be undertaken at the screening visit if no previous biopsy confirmation available.

And;

* Having failed steroids (topical, intralesional, systemic) and are candidates for antimalarial therapy
* Negative ANA

Have no history of latent or active TB prior to screening.

Exclusion Criteria:

* Subjects allergic to sunscreens
* Prior treatment with anti-TNF therapies
* Subjects who do not have a previous skin biopsy result confirming a DLE diagnosis and who are unwilling to undergo this procedure at screening.
* Subjects currently receiving systemic steroid therapy (or have received in the last 3 months)
* Known hypersensitivity to Enbrel® (etanercept) or any of its components or known to have antibodies to etanercept.
* Prior or concurrent use of cyclophosphamide therapy
* Concurrent sulfasalazine therapy.
* Known HIV-positive status or known history of any other immuno-suppressing disease.
* Any mycobacterial disease or high risk factors for tuberculosis (TB), such as family member with TB, positive purified protein derivative (PPD) or taking anti-tuberculosis medication
* Active or chronic infection within 4 weeks before screening visit, or between the screening and baseline visits.
* Severe comorbidities (diabetes mellitus requiring insulin; CHF of any severity; or myocardial infarction, cerebrovascular accident or transient ischemic attack within 6 months of screening visit; unstable angina pectoris; uncontrolled hypertension (sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg); oxygen-dependent severe pulmonary disease; history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma of the skin or in situ cervical cancer])
* Systemic lupus erythematosus, history of multiple sclerosis, transverse myelitis, optic neuritis or seizure disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients responding to study treatment using the Cutaneous Lupus Erythematous Disease Area Severity Index(CLASI)defined as a decrease of 50% form baseline. | 20 weeks

SECONDARY OUTCOMES:
Change from baseline to week 20 in Dermatology Life Quality Index and Pysician's Global Assessment of disease measurements | 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Dermatology Centers, Miami, Florida, United States